CLINICAL TRIAL: NCT01848639
Title: ALdosterone Antagonist Chronic HEModialysis Interventional Survival Trial (ALCHEMIST), Phase III b
Brief Title: ALdosterone Antagonist Chronic HEModialysis Interventional Survival Trial
Acronym: ALCHEMIST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Collaborators: Central Hospital, Nancy, France (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ALCHEMIST; RB 12-079 (Other: CHRU Brest)
Record Dates: First submitted 2013-05-03; First posted 2013-05-07 (Estimated); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: End Stage Renal Failure on Dialysis
Keywords: chronic kidney disease; end-stage renal disease; hemodialysis (ESRD); cardiovascular morbimortality; aldosterone antagonist; spironolactone
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic | interventions — Spironolactone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Spironolactone (Active Comparator): After a month in run-in period under 25 mg per 2 days of spironolactone administered per os in practice after dialysis session three times a week, patients will be randomized to spironolactone. The dose should be increased to 25 mg once daily and could be adjusted in using an algorithm used in the EPHESUS and EMPHASIS-HF trials.
  Interventions: Drug: Spironolactone
- Placebo (Placebo Comparator): After a month in run-in period under 25 mg per 2 days of spironolactone administered per os in practice after dialysis session three times a week, patients will be randomized to placebo. The dose should be increased to 25 mg once daily and could be adjusted in using an algorithm used in the EPHESUS and EMPHASIS-HF trials.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Spironolactone — After a month in run-in period under 25 mg per 2 days of spironolactone administered per os in practice after dialysis session three times a week, patients will be randomized to spironolactone. The dose should be increased to 25 mg once daily and could be adjusted in using an algorithm used in the EPHESUS and EMPHASIS-HF trials.
  Arms: Spironolactone
Drug: Placebo — After a month in run-in period under 25 mg per 2 days of spironolactone administered per os in practice after dialysis session three times a week, patients will be randomized to placebo. The dose should be increased to 25 mg once daily and could be adjusted in using an algorithm used in the EPHESUS and EMPHASIS-HF trials.
  Arms: Placebo

SUMMARY:
This study is designed to etablish the effects of spironolactone in comparison to placebo on the composite endpoint of nonfatal Myocardial Infarction (MI) and acute coronary syndrome, hospitalization for heart failure, nonfatal stroke or cardiovascular-induced death. The primary endpoint will be the time to onset of the first incident.

DETAILED DESCRIPTION:
* During a run-in period : Spironolactone will be initially administered per os at a 25 mg dose per two days in practice after the session, three times per week
* Patients will be randomized (spironolactone vs. placebo) and titrated over one month to a maximum single dose of 25 mg/d
* However if kalemia is greater than or equal to 5.5 mmol / l twice on this run-in period or on the day of randomization, patient won't be randomized.
* A pre-specified algorithm for the management of the risk of incident hyperkalemia will be followed, including dose adjustment, temporary cessation of study treatment, in addition to usual dietary measures and the use of chelating resins and low-potassium dialysis baths
* Patients will be followed for a mean of 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Adult men and women on HD for at least 45 days for ESRD regardless of the etiology including diabetes, with at least 3 HD sessions per week
* Presenting at least one of the follow comorbidities, cardiovascular abnormalities or CV risk factors:
* Left ventricular hypertrophy defined by left ventricular mass > 130 g/m2 in men and 100 g/m2 in women (echocardiography)
* OR Cornell (RaVL + SV3) >28 mm in men, > 20 mm in women(ECG)
* OR left ventricular ejection fraction < 40%
* OR large QRS > 0.14 sec
* OR Left bundle branch block (ECG) measured during the twelve months preceding inclusion; diabetes;
* OR history of cardiovascular disease: coronary artery disease, symptomatic lower limb peripheral arterial disease, carotid or renal artery stenosis > 50%, stroke, hospitalization for heart failure, permanent atrial fibrillation (AF), oral anticoagulant treatment for AF, valvular heart prosthesis,
* OR CRP > 5 mg/l for 3 months without infectious or neoplastic disease documented in progress

Exclusion Criteria:

* history of hypersensitivity to spironolactone or galactose intolerance
* the Lapp lactase deficiency or malabsorption of glucose or galactose
* hyperkalemia > 5.5 mmol/l during the two weeks prior to enrolment
* history of unscheduled hemodialysis for hyperkalemia during the last six months
* hospitalization for hyperkalemia during the last six months
* patients with imperative indication of a combination of ACEI and sartan or renin inhibitor (each being authorized separately), NSAIDS, Cox-2 inhibitors
* kidney transplant scheduled within the year
* symptomatic interdialytic hypotension
* acute systemic disease
* uncompensated hypothyroidism
* acute hyperthyroidism
* any prior or concomitant clinical condition compromising the inclusion, in the discretion of the investigator
* cardiac transplant
* severe uncontrolled arrhythmia
* stroke within 3 months prior to enrolment
* acute coronary syndrome in the previous month inclusion
* recent (1 month) or planned coronary revascularization by angioplasty
* recent (3 months) or planned cardiovascular surgery (excluding HD vascular access)
* non menopausal women or without effective contraceptive methods
* pregnancy, breastfeeding or planning a pregnancy within 2 years
* non compliance
* protected adult
* SBP > 200 mmHg and/or DBP > 110 mmHg
* Concomitant treatment can not be stopped by another potassium-sparing diuretic, a potassium supplements, AINS or Cox 2 inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 823 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2022-11 (Actual); Study Completion 2022-11 (Actual)

PRIMARY OUTCOMES:
The time to onset of the first incident :non-fatal MI or acute coronary syndrome or hospitalization for heart failure or nonfatal stroke or cardiovascular (CV) death | 25 months

SECONDARY OUTCOMES:
Determine the effects of spironolactone compared to placebo on the composite winratio endpoint | 24 months
  Following a hierarchical strategy of statistical tests including the primary endpoint.
  Composite winratio endpoint of: all-cause mortality at 2 years according to the Finkelstein and Schoenfeld method.
Determine the effects of spironolactone compared to placebo on the composite winratio endpoint | 24 months
  Following a hierarchical strategy of statistical tests including the primary endpoint.
  Composite winratio endpoint of: time until a cardiovascular event (hospitalization for heart failure, or non-fatal myocardial infarction, or acute coronary syndrome or non-fatal stroke) at 2 years according to the Finkelstein and Schoenfeld method.
non-cardiovascular mortality rate | 24 months
  Additional secondary objectives will be considered in the context of hypothesis generation
cumulative accident rates forming the primary endpoint | 24 months
  Additional secondary objectives will be considered in the context of hypothesis generation
The time of survival without a major CV event (non fatal MI, acute coronary syndrome, hospitalization for heart failure, non-fatal stroke, cardiac arrest resuscitation) | 24 months
  Additional secondary objectives will be considered in the context of hypothesis generation
Incidence of procedures related to stenosis or vascular access thrombosis for hemodialysis (HD) | 24 months
  Additional secondary objectives will be considered in the context of hypothesis generation
Incidence of coronary or peripheral revascularizations (including lower limb amputations) | 24 months
  Additional secondary objectives will be considered in the context of hypothesis generation
Blood pressure (systolic and diastolic pressure) | 24 months
  Additional secondary objectives will be considered in the context of hypothesis generation
Blood pressure's variability inter visit (systolic and diastolic pressure) | 24 months
  Additional secondary objectives will be considered in the context of hypothesis generation
The occurrence of atrial fibrillation | 24 months
  Additional secondary objectives will be considered in the context of hypothesis generation
Incidence of hyperkalemia> 6 mmol/l | 24 months
  Additional secondary objectives will be considered in the context of hypothesis generation
Estimation of the effect of treatment on quality of life. | 24 months
  KDQoL questionnaire ; minimum value = 0 ; maximum value = 100 ; higher score means a better outcome
Estimation of the effect of treatment on quality of life. | 24 months
  Minnesota questionnaire ; minimum value = 0 ; maximum value = 100 ; higher score means a better outcome
Estimation of the effect of treatment on quality of life. | 24 months
  SF36 questionnaire ; minimum value = 0 ; maximum value = 100 ; higher score means a better outcome

OTHER OUTCOMES:
Ancillary study:establishment of a biological collection (serum bank and DNA biobank) for future biomarker studies | 24 months
Ancillary study:morbimortality data | 3, 5 and 10 years of follow-up after the double-blind study

CONTACTS AND LOCATIONS:
Locations (70):
- Hôpital Erasme- Bruxelles, Brussels, Belgium
- France (68):
  - CH Ardeche Nord, Annonay, Ardeche
  - CHU Amiens, Amiens
  - CH Avignon, Avignon
  - CHU Besançon, Besançon
  - CH Boulogne Sur Mer, Boulogne-sur-Mer
  - CHRU Brest, Brest
  - CHU Caen, Caen
  - CH Cahors, Cahors
  - CH Chambéry, Chambéry
  - CHPC Cherbourg, Cherbourg
  - AURAL Colmar, Colmar
  - Hopitaux Civils de Colmar, Colmar
  - APHP Henri Mondor, Créteil
  - CHU Dijon Hôpital du Bocage, Dijon
  - AGDUC Grenoble, Grenoble
  - AURAL Haguenau, Haguenau
  - CH Haguenau, Haguenau
  - La Roche Sur Yon, La Roche-sur-Yon
  - Polyclinique de Lagny, Lagny
  - Clinique Lille, Lille
  - CHU Lille, Lille
  - ALURAD Limoges, Limoges
  - CHU Limoges, Limoges
  - CHU de Lyon, Lyon
  - AURAL La Croix Rousse, Lyon
  - CH St Joseph-St Luc, Lyon
  - AURAL Lyon, Lyon
  - Clinique Bouchard, Marseille
  - Adpc Marseille, Marseille
  - APHM Marseille, Marseille
  - Association de Metz, Metz
  - ALTIR Metz, Metz
  - CHR Metz-Thionville, Metz
  - AURAL Mulhouse, Mulhouse
  - CH Mulhouse, Mulhouse
  - CHU Nancy, Nancy
  - CHU Nantes, Nantes
  - CHU Nice, Nice
  - Clinique St Georges, Nice
  - AP-HP La Salpêtrière, Paris
  - AURA Paris 14ème, Paris
  - AURA Paris Plaisance, Paris
  - Hôpital Tenon, Paris
  - AP-HP Necker, Paris
  - Institut Mutualiste Montsouris, Paris
  - CHU Lyon Sud, Pierre-Bénite
  - CHU de Reims, Reims
  - ARPDD Reims, Reims
  - CHU Rennes, Rennes
  - ECHO Confluent, Rezé
  - Centre de Perharidy, Roscoff
  - CH Roubaix, Roubaix
  - CHG St Brieuc, Saint-Brieuc
  - CHU de la Réunion Hôpital Félix Guyon, Saint-Denis
  - Aub Saint Malo, St-Malo
  - Ch Saint Malo, St-Malo
  - AURAL St Anne (AURAL Strasbourg), Strasbourg
  - CHU Strasbourg, Strasbourg
  - Clinique Sainte Anne, Strasbourg
  - AURAL Strasbourg, Strasbourg
  - CHU Toulouse, Toulouse
  - CHU Tours, Tours
  - CH Troyes, Troyes
  - CH Valenciennes, Valenciennes
  - ALTIR Nancy, Vandœuvre-lès-Nancy
  - Hôpitaux Privés de Metz- Hôpital Robert Schuman, Vantoux
  - CH Verdun, Verdun
  - CH Vichy, Vichy
- CH Princesse Grace, Monaco, Monaco

IPD SHARING:
Plan to Share IPD: Yes
Statistical Analysis Plan
Supporting Information: SAP
URL: https://cic-p-nancy.fr/wp-content/uploads/2023/10/Alchemist_SAP-V3-and-SAP-QoL-V08-20231005-signe.pdf

REFERENCES:
- [Derived] Rossignol P, Zannad F, Massy Z, Azizi M, Chorfa F, Coadic J, Ferreira JP, Saraiva F, Mottier D, Guillemin F, Ngueyon Sime W, Bouali S, Rossignol B, Nortier J, Simon I, Robino C, Davin M, Bataille PM, Chantrel F, Castin N, Esnault V, Kazes I, Hannedouche T, Kamar N, Achard JM, Fenerol C, Achard-Hottelart C, Dimitrov Y, Girerd N, Maucort-Boulch D, Frimat L; ALCHEMIST study group. Spironolactone in patients on chronic haemodialysis at high risk of adverse cardiovascular outcomes (ALCHEMIST): a multicentre, double-blind, randomised, placebo-controlled trial and updated meta-analysis. Lancet. 2025 Aug 16;406(10504):705-718. doi: 10.1016/S0140-6736(25)01194-8. PMID 40818851
- [Derived] Hasegawa T, Nishiwaki H, Ota E, Levack WM, Noma H. Aldosterone antagonists for people with chronic kidney disease requiring dialysis. Cochrane Database Syst Rev. 2021 Feb 15;2(2):CD013109. doi: 10.1002/14651858.CD013109.pub2. PMID 33586138